CLINICAL TRIAL: NCT03049956
Title: Diagnostic Accuracy of Repetitive Ocular Vestibular Evoked Myogenic Potentials in Myasthenia Gravis (OMG Study)
Brief Title: OVEMP in Myasthenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Konrad Peter Weber, PD Dr.med., University of Zurich
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: 2016-01109
Record Dates: First submitted 2017-02-01; First posted 2017-02-10 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Myasthenia Gravis, Ocular
Keywords: Ocular Vestibular Evoked Myogenic Potentials
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Masking Description: Blinded diagnostic accuracy study (index test vs. reference standard).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with clinical suspicion of ocular myasthenia gravis (Experimental)
  Interventions: Diagnostic Test: Ocular vestibular evoced myogenic potentials

INTERVENTIONS:
Diagnostic Test: Ocular vestibular evoced myogenic potentials — The oVEMP technique is an accepted standard for testing otolith function in vestibular patients. It represents a quick, simple and non-invasive technique utilizing repetitive stimulation of the otolith organs with bone-conducted vibration to elicit an extraocular muscle response. Repetitive oVEMP stimulation leads to a characteristic decrement in patients with myasthenia, which can be quantified with surface electromyography from the inferior oblique muscle underneath the eye.

SUMMARY:
Myasthenia gravis is an autoimmune disorder of neuromuscular transmission, characterized by fluctuating muscle weakness and fatigability. In isolated ocular myasthenia, when only the extraocular muscles are involved, most common ancillary tests, such as acetylcholine receptor autoantibodies and repetitive nerve stimulation, are often negative.

A simple, quick and non-invasive test for ocular myasthenia based on ocular vestibular evoked myogenic potentials (oVEMP) was recently developed.

The main goal of the study is to validate repetitive oVEMP stimulation in a blinded diagnostic accuracy study in order to facilitate early and accurate diagnosis of ocular myasthenia.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Patients with diplopia and/or ptosis suspicious for myasthenia gravis.

Exclusion Criteria:

* Vestibular disorders
* Significant systemic myasthenia symptoms (respiration or swallowing difficulties) unable to undergo oVEMP testing.
* Patients with significant cardiac or respiratory disease will be excluded from the Tensilon test as part of the reference standard.
* Women who are pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Decrement (as quantified in %) of repetitive 20 Hz ocular vestibular-evoked myogenic potentials (oVEMP) | The primary outcome measure (index test oVEMP) will be assessed at baseline, in conjunction with reference standard/standard clinical workup (including blood analysis, neurological exam, edrophonium test, electromyography, single-fiber electromyography).
  oVEMP have been established as a standard clinical test of otolith function. Based on this technique, repetitive oVEMP stimulation, as a novel method for detecting ocular myasthenia gravis, was recently developed. Using this method, a response decrement in extraocular muscles can be quantified. The method is based on the conventional oVEMP montage with surface electrodes placed below the eyes. In order to elicit a response decrement, trains of ten bone-conducted vibration bursts at repetition rates of 20Hz will be applied with a hand-held 'minishaker' to the forehead. The oVEMP in response to these repetitive vibration stimuli will be measured in sustained upgaze from both inferior oblique muscles via surface electrodes. The magnitude of the decrement will be calculated as the difference between the amplitude of the second stimulus repetition and the mean amplitude of the fifth to ninth stimulus repetition. For further Information see: Valko et al. 2016 PMID:26791146

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Ophthalmology/Neurology Department, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valko Y, Rosengren SM, Jung HH, Straumann D, Landau K, Weber KP. Ocular vestibular evoked myogenic potentials as a test for myasthenia gravis. Neurology. 2016 Feb 16;86(7):660-8. doi: 10.1212/WNL.0000000000002383. Epub 2016 Jan 20. PMID 26791146
- [Derived] Handzic A, Furter MP, Messmer BC, Wirth MA, Valko Y, Fierz FC, Margolin EA, Weber KP. Multivariable Prediction Model for Suspected Ocular Myasthenia Gravis: Development and Validation. J Neuroophthalmol. 2025 Apr 21. doi: 10.1097/WNO.0000000000002346. Online ahead of print. PMID 40257852
- [Derived] Valko Y, Wirth MA, Fierz FC, Schesny MK, Rosengren S, Schmuckle-Meier T, Bockisch CJ, Straumann D, Schreiner B, Weber KP. Accuracy of Repetitive Ocular Vestibular-Evoked Myogenic Potentials to Diagnose Myasthenia Gravis in Patients With Ptosis or Diplopia. Neurology. 2024 May;102(10):e209395. doi: 10.1212/WNL.0000000000209395. Epub 2024 Apr 26. PMID 38669629